CLINICAL TRIAL: NCT02386774
Title: Innovative Imaging of the Conjunctiva, Cornea, and Ocular Adnexa : Study of a Handheld in Vivo Confocal Microscope and of a Fluorescent in Vivo Confocal Microscope
Brief Title: Innovative Imaging of the Conjunctiva, Cornea, and Ocular Adnexa
Acronym: INNOV-EYE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1208180; 2015-A00331-48 (Other: ANSM)
Record Dates: First submitted 2015-02-20; First posted 2015-03-12 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Corneal Disease; Blepharitis; Lacrimal Apparatus Diseases
Keywords: In vivo confocal microscopy; corneal disease; Blepharitis; Lacrimal Apparatus Diseases; Microscopy, Confocal
MeSH Terms: conditions — Corneal Diseases; Blepharitis; Lacrimal Apparatus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- an ocular or ocular adnexa disease (Other): patient presenting with an ocular or ocular adnexa disease in the Dermatology or Ophthalmology ward.
  Interventions: Device: Handheld IVCM Vivascope 3000 (Caliber/Mavig) anesthesic eyedrop : oxybuprocaïne Thea 1,6 mg/0,4 ml; Device: Multifluorescence IVCM vivascope 1500 ML (Caliber/Mavig); Procedure: microangiography
- diabetic patients (Other)
  Interventions: Device: Multifluorescence IVCM vivascope 1500 ML (Caliber/Mavig); Procedure: microangiography

INTERVENTIONS:
Device: Handheld IVCM Vivascope 3000 (Caliber/Mavig) anesthesic eyedrop : oxybuprocaïne Thea 1,6 mg/0,4 ml — used anesthesic eyedrop : oxybuprocaïne Thea 1,6 mg/0,4 ml
  Arms: an ocular or ocular adnexa disease
Device: Multifluorescence IVCM vivascope 1500 ML (Caliber/Mavig) — used for Multifluorescence IVCM
  * anesthesic eyedrop : oxybuprocaïne (1,6 mg/0,4 ml)
  * Fluorescein 0,5%, Rose Bengal , Infracyanine
Procedure: microangiography — realization of the microangiography with intravenous injection of fluoresceine and indocyanine green.

SUMMARY:
In vivo confocal microscopy (IVCM) used in tertiary care ophthalmology centers is performed with two reflectance microscopes attached on a mounting with limited movement along the XYZ axes. Consequently, ocular diseases in the central area have been described (mostly cornea and adjacent conjunctiva). Two dermatology IVCM (an handheld small IVCM and a multifluorescent one) present significant innovations that the investigators want to assess in ophthalmology for the diagnosis of conjunctiva, cornea, eyelid and lachrymal tract diseases. The handheld IVCM have unlimited degrees of freedom and a small diameter objective. It could dramatically increase the area accessible to IVCM (whole conjunctiva, eyelids, proximal lachrymal tract) (part 1 of the present study). The fluorescent IVCM allows the use of a wide range of fluorescent markers liable to increase the specificity of the diagnosis by revealing staining patterns corresponding to a specific disease and not to others (part 2 of the study)

ELIGIBILITY:
Inclusion Criteria:

* Presenting with an ocular or ocular adnexa disease (infectious keratitis, stromal dystrophy, corneal surgery, ocular surface toxicity of eyedrops, cornea-conjunctival tumors, chronic blepharitis, eyelid tumors, diseases of the proximal lachrymal tract).
* For the microangiography: diabetic patients

Exclusion Criteria:

* Allergy to one of the 3 dyes (fluorescein, indocyanine green, rose Bengal)
* Pregnancy and breast feeding
* Predicable impossible follow up
* For patient volunteer for intravenous injections: beta blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance (sensitivity (se) and specificity (sp)) of the handheld IVCM in ocular surface and adnexa diseases | 1 year

SECONDARY OUTCOMES:
handheld IVCM : sensitivity (se) and specificity (sp) in each 8 subgroups of diseases | 1 year
handheld IVCM : positive and negative predictive values in each 8 subgroups of diseases | 1 year
handheld IVCM : AUC of the ROC curve in each 8 subgroups of diseases | 1 year
handheld IVCM : factors influencing image quality | 1 year
  using a scale to 3 levels (2 : optic diagnosis ; 1 : presence of artifacts but possible optic diagnosis ; 0 :impossible optic diagnosis)
handheld IVCM : determining the limits of the tumor | 1 year
  (in the particular case of tumors requiring surgery)
fluorescence : staining patterns obtained for each disease group | 1 year
fluorescence : characteristics of the micro-angiography | 1 year
  characteristics of the conjunctival vessels in normal and diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Gilles THURET, MD PhD, Principal Investigator — CHU de St Etienne
Locations (2):
- France (2):
  - Chu de Saint Etienne, Saint-Etienne, Dermatology
  - Chu de Saint Etienne, Saint-Etienne, Ophtalmology

IPD SHARING:
Plan to Share IPD: No